CLINICAL TRIAL: NCT03010488
Title: Are Bright Lights and Regulated Sleep Effective Treatment for Depression.
Brief Title: Are Bright Lights and Regulated Sleep Effective Treatment for Depression?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, David J. Hellerstein, Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7361; 7361 (Other: IRB)
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Sleep Phase Rhythm Disturbance; Sleep Deprivation
Keywords: Chronotherapy; Light Therapy
MeSH Terms: conditions — Sleep Deprivation | interventions — Phototherapy; Sleep Phase Chronotherapy; Eye Protective Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid Sleep Shift (Experimental): Assigned Sleep Times designed to shift sleep times over several days from Baseline to desired through morning light therapy while wearing goggles.
  Interventions: Behavioral: Morning Light Therapy; Behavioral: Assigned Sleep Times; Device: Goggles
- Gradual Sleep Shift (Active Comparator): Assigned Sleep Times designed gradually shift sleep from current to desired sleep times while using morning light therapy while wearing goggles.
  Interventions: Behavioral: Morning Light Therapy; Behavioral: Assigned Sleep Times; Device: Goggles

INTERVENTIONS:
Behavioral: Morning Light Therapy — 10,000 Lux light for 30 minutes through a light box each morning at patient's desired wake up time.
  Other Names: Light Therapy
Behavioral: Assigned Sleep Times — Sleep times will be assigned to subjects that will allow them to drive their regular sleep times closer to those they determine to be optimal at study initiation.
  Other Names: Sleep Phase Advance
Device: Goggles — Subjects will wear goggles during saliva collection and Bright Light Therapy

SUMMARY:
Previous data suggest some depressed patients act as if their internal biological clock is out of sync with the outside world and re-aligning their clock with the timing of sunlight lessens their depressed mood and accompanying depressive symptoms. This "chronotherapy" may produce remission during the first week of treatment while causing minimal problems. This study aims to demonstrate the efficacy of chronotherapy by comparing two protocols for inducing sleep phase advance. Which chronotherapy condition a participant will receive will be determined randomly (i.e., by chance, essentially a computerized flip of a coin). Prior to determination of which protocol a patient will follow, each patient will declare their desired sleep time (for example, 11 p.m. to 7 a.m.). All patients will be assigned specific times to sleep and sit in front of bight lights wearing clear or amber goggles. Assigned sleep times will differ between groups using different strategies to shift the timing of their sleep from their ideal sleep time as determined by their Morningness-Eveningness Questionnaire (MEQ) score to their desired sleep time. All participants will be rated daily by telephone for the first week following randomization, and then weekly for an additional five weeks. Whenever possible, weekly visits will be in person, although telephone visits will be allowed. All participants will be rated at baseline, 1 week and 6 weeks by an Independent Evaluator blind to treatment assignment (as well as the nature of the treatment and if it has occurred or not). After the six week post-randomization evaluation, all participants will be offered six months of continued treatment and be rated monthly. Treatment during this six month period may consist of Chronotherapy or conventional antidepressants as the patient and doctor determine. Standard ratings of depression, over-all illness and functioning will be obtained. Change in the symptom measures will determine treatment efficacy. Analysis of saliva melatonin levels, sleep logs and activity monitor data will measure the timing of the biological clock and whether it has been shifted by the treatment. Measures of functioning will determine whether functioning improves coincident with, independent of, or subsequent to mood improvement.

DETAILED DESCRIPTION:
This study will investigate the utility of regimented sleep and lights in depressed subjects. Based on current timing of sleep, desired sleep time and responses to the Morningness-Eveningness Questionnaire, each subject who remains significantly depressed at their randomization (usually 2nd) visit, will be randomly assigned to one of two regimented sleep and light use protocols. On the night beginning their assigned regimented protocol, each subject will wear amber goggles for five hours and collect half hourly saliva samples for four hours. Each morning they will sit in front of a light box wearing goggles. During the first week following the start of the regimented protocol, they will complete self-report forms and have a telephone interview to document their depressive symptoms. They will have weekly in person interviews for six weeks and evaluations by an independent evaluator in person or by telephone at randomization, 2 and 6 weeks. Prior to their Week 2 Visit, they will wear the goggles for the four hours prior to their assigned bedtime and for the three hours prior to their assigned bedtime, they will collect half hourly saliva samples. At their Week 6 interview, they and their doctor will determine whether they have improved sufficiently or not. Their doctor will discuss with them whether it makes sense for them to continue the same regimented sleep/light schedule, make a change to it or switch to or add additional treatment, such as antidepressant medication. They will then be followed with study ratings monthly for six months, during which treatment is unrestricted; that is, the doctor and patient can determine what the treatment during this time will be. Following the six months follow-up, a referral will be made if appropriate.

All saliva samples will be analyzed for melatonin concentration.

ELIGIBILITY:
Inclusion Criteria:

* Currently Depressed
* In reasonably good physical health

Exclusion Criteria:

* Bipolar Disorder (I, II, or unspecified)
* History of psychosis
* Unstable medical condition
* Current (past 6 months) drug or alcohol use disorder
* Need for hospitalization
* Treating clinician determines not to include patient in this protocol
* Currently taking medications approved for the treatment of depression
* Un- or poorly controlled hypertension
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-11; Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Stewart, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Depression Evaluation Service - New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All non-identifiable data will be made available to qualified researchers on request to the study PI.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Information will be sent as soon as is practical and will be available as long as the PI is available.
Access Criteria: Legitimate research agenda, including but not limited to request to double-check presented or published results and novel analyses.

RESULTS

PARTICIPANT FLOW:
Groups:
- Rapid Sleep Shift: Assigned Sleep Times designed to shift sleep times over several days from Baseline to desired through morning light therapy while wearing clear goggles.
  Morning Light Therapy: 10,000 Lux light for 30 minutes through a light box each morning at patient's desired wake up time.
  Assigned Sleep Times: Sleep times will be assigned to subjects that will allow them to drive their regular sleep times closer to those they determine to be optimal at study initiation.
  Goggles: Subjects will wear goggles during saliva collection and Bright Light Therapy
- Gradual Sleep Shift: Assigned Sleep Times designed gradually shift sleep from current to desired sleep times while using morning light therapy while wearing amber (blue blocking) goggles.
  Morning Light Therapy: 10,000 Lux light for 30 minutes through a light box each morning at patient's desired wake up time.
  Assigned Sleep Times: Sleep times will be assigned to subjects that will allow them to drive their regular sleep times closer to those they determine to be optimal at study initiation.
  Goggles: Subjects will wear goggles during saliva collection and Bright Light Therapy
Period: Overall Study
Arm/Group | Rapid Sleep Shift | Gradual Sleep Shift
Started | 22 | 22
Completed | 17 | 15
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapid Sleep Shift | Gradual Sleep Shift | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (14.3) | 38.8 (16.4) | 38.3 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 17 | 17 | 34
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: 17-Item Hamilton Rating Scale for Depression Score (Independent Evaluator)
Description: Independent Evaluator's Week 6 17-item Hamilton Rating Scale for Depression Summary Score. The 17-item Hamilton is the standard measure of depression severity for clinical trials of antidepressants and was chosen as the primary outcome measure over other depression rating scales to ensure compatibility of study results with our meta-analyses and ongoing studies of expectancy. Although the Hamilton list 24 items, the scoring is based on both the first 17 items and the full 24 items.
  sum of the scores of the first 17 items (range from 0 to 54): 0-7 = NORMAL 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression >=23 = Very Severe Depression
Time Frame: Week 6
Population: Due to rater availability we weren't able to get independent evaluations on all participants. The numbers listed or the number we were able to get independent evaluations on.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rapid Sleep Shift | Gradual Sleep Shift
Number analyzed (Participants) | 18 | 15
units on a scale | 8.66 (6.09) | 10.46 (7.79)

2. Secondary Outcome: Participant Sleep Efficiency
Description: Sleep Efficiency (percentage of time spent sleeping during target sleep period) as measured by activity monitor and sleep logs.
  Sleep logs: Patients were instructed to record all sleep periods in the daily log by marking boxes representing 15-minute intervals. They were also requested to wear the Actigraph activity monitor at all times except for bathing, swimming, or any other activities requiring immersion of the wrist. In addition, patients were provided with schedules delineating their allowed sleep time each day.
  Patients chose their target sleep times (an eight-hour time they desired their sleep to occur) and completed the Morningness-Eveningness Questionnaire (MEQ) to estimate the timing of their circadian clocks, including ideal sleep and wake-up times.
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Rapid Sleep Shift | Gradual Sleep Shift
Number analyzed (Participants) | 7 | 7
percentage of time | 76.43 (10.82) | 68.23 (28.27)

ADVERSE EVENTS:
Time Frame: 7.5 months
Arm/Group | Rapid Sleep Shift | Gradual Sleep Shift
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Informed Consent Form (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT03010488/ICF_000.pdf
  • Study Protocol (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03010488/Prot_001.pdf
  • Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03010488/SAP_002.pdf